CLINICAL TRIAL: NCT03200093
Title: Secondary Prophylaxis With Oral Vancomycin for Clostridium Difficile Recurrence: A Randomized Control Study
Brief Title: Oral Vancomycin for Preventing Clostridium Difficile Recurrence
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment due to few eligible participants.
Sponsor: Rochester General Hospital (Other)
Responsible Party: Principal Investigator, Maryrose R Laguio-Vila, Physician, Rochester General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIC 1745-B-17 Laguio-Vila
Record Dates: First submitted 2017-06-23; First posted 2017-06-27 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; C diff; Oral Vancomycin; Prophylaxis
MeSH Terms: conditions — Clostridium Infections | interventions — Vancomycin; Drug Evaluation

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After enrollment, study pharmacists will randomize the participants to receive either oral vancomycin or placebo. Participants, care providers, investigators, and outcomes assessors will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral vancomycin (Experimental): Oral vancomycin solution 125 mg in 2.5 mL, combined with 2.5 ml Ora-Sweet solution, to total 5 mL.
  Taken by mouth once daily for:
  1. If the total duration of systemic antibiotics is less than or equal to 14 days, oral vancomycin will be taken for the duration of the systemic antibiotics plus three days.
  2. If the total duration of systemic antibiotics is greater than 14 days, oral vancomycin will be taken for the duration of the systemic antibiotics plus seven days.
  Interventions: Drug: Oral Vancomycin
- Placebo arm (Placebo Comparator): Ora-Sweet 5 mL
  Taken by mouth once daily for:
  1. If the total duration of systemic antibiotics is less than or equal to 14 days, placebo will be taken for the duration of the systemic antibiotics plus three days.
  2. If the total duration of systemic antibiotics is greater than 14 days, placebo will be taken for the duration of the systemic antibiotics plus seven days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Vancomycin — Oral vancomycin solution 125 mg in 2.5 mL combined with 2.5 mL Ora-Sweet. A total of 5 mL combined solution taken by mouth once daily.
  Other Names: Study drug
  Arms: Oral vancomycin
Drug: Placebo — Ora-Sweet 5mL taken by mouth once daily.
  Other Names: Study placebo
  Arms: Placebo arm

SUMMARY:
This study evaluates the role of oral vancomycin in the prevention of recurrent Clostridium difficile for hospitalized patients receiving systemic antibiotic therapy. Half of participants will receive oral vancomycin daily, while the other half will receive a placebo.

DETAILED DESCRIPTION:
Clostridium difficile colitis is a significant cause of morbidity and mortality among hospitalized patients. Following the first episode, up to 15% of people experience recurrent disease. A major risk factor for recurrent disease is exposure to systemic antibiotics.

Oral vancomycin given four times daily is one of the treatments for Clostridium difficile infection; it is not known if giving oral vancomycin at a lower dose such as once daily may help prevent recurrences. Oral vancomycin may be most helpful in preventing recurrences when given to patients at greatest risk of recurrent disease, such as when they are receiving systemic antibiotics.

To evaluate this, the investigators propose comparing the rates of recurrent Clostridium difficile infection in patients who receive oral vancomycin with systemic antibiotics to when patients take systemic antibiotics alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Any history of Clostridium difficile infection based on a positive Clostridium difficile stool test performed at a lab affiliated with Rochester Regional Health System or patient report
* A new in-patient admission, with an antibiotic treatment plan for greater than 48 hours

Exclusion Criteria:

* Documented allergy and/or adverse drug reaction to vancomycin
* Pregnant
* Patients who are admitted with a current episode of Clostridium difficile infection
* Patients with total colectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
30-day recurrent Clostridium difficile infection | 30 days
  A positive Clostridium difficile stool test in the 30 days following completion of the systemic antibiotic treatment.

SECONDARY OUTCOMES:
90-day recurrent Clostridium difficile infection | 90 days
  A positive Clostridium difficile stool test in the 90 days following completion of the systemic antibiotic treatment.
30-day hospital re-admission | 30 days
  All-cause re-admission to any hospital
30-day mortality | 30 days
  All-cause mortality in the 30 days following completion of the systemic antibiotics

OTHER OUTCOMES:
Impact of duration of systemic antibiotics on Clostridium difficile recurrence | 90 days
  Comparing the frequency of a positive Clostridium difficile stool test in the 90 days following completion of systemic antibiotics, when the duration of systemic antibiotics was less than or equal to 14 days compared to longer durations.
Impact of acid-suppressing medications on Clostridium difficile recurrence | 90 days
  Comparing the frequency of a positive Clostridium difficile stool test in the 90 days following completion of systemic antibiotics, when the participant was receiving acid-suppressing medications compared to those on none.
Impact of age on Clostridium difficile recurrence | 90 days
  Comparing the frequency of a positive Clostridium difficile stool test in the 90 days following completion of systemic antibiotics, when the participant was older than 65 years of age compared to younger.
Impact of systemic antibiotic class on Clostridium difficile recurrence | 90 days
  Comparing the frequency of a positive Clostridium difficile stool test in the 90 days following completion of systemic antibiotics, when the participant was receiving systemic antibiotics considered "high risk" for Clostridium difficile compared to those taking "low risk" antibiotics.
Vancomycin resistance isolated | 90 days
  Isolation of a vancomycin-resistant bacteria during an infectious workup, if clinically indicated

CONTACTS AND LOCATIONS:
Overall Officials: Maryrose R Laguio-Vila, MD, Principal Investigator — Rochester General Hospital
Locations (1):
- Rochester General Hospital, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lessa FC, Mu Y, Bamberg WM, Beldavs ZG, Dumyati GK, Dunn JR, Farley MM, Holzbauer SM, Meek JI, Phipps EC, Wilson LE, Winston LG, Cohen JA, Limbago BM, Fridkin SK, Gerding DN, McDonald LC. Burden of Clostridium difficile infection in the United States. N Engl J Med. 2015 Feb 26;372(9):825-34. doi: 10.1056/NEJMoa1408913. PMID 25714160
- [Background] Surawicz CM, Brandt LJ, Binion DG, Ananthakrishnan AN, Curry SR, Gilligan PH, McFarland LV, Mellow M, Zuckerbraun BS. Guidelines for diagnosis, treatment, and prevention of Clostridium difficile infections. Am J Gastroenterol. 2013 Apr;108(4):478-98; quiz 499. doi: 10.1038/ajg.2013.4. Epub 2013 Feb 26. PMID 23439232
- [Background] Gupta A, Khanna S. Community-acquired Clostridium difficile infection: an increasing public health threat. Infect Drug Resist. 2014 Mar 17;7:63-72. doi: 10.2147/IDR.S46780. eCollection 2014. PMID 24669194
- [Background] Vincent C, Manges AR. Antimicrobial Use, Human Gut Microbiota and Clostridium difficile Colonization and Infection. Antibiotics (Basel). 2015 Jul 3;4(3):230-53. doi: 10.3390/antibiotics4030230. PMID 27025623
- [Background] Brandt LJ, Aroniadis OC, Mellow M, Kanatzar A, Kelly C, Park T, Stollman N, Rohlke F, Surawicz C. Long-term follow-up of colonoscopic fecal microbiota transplant for recurrent Clostridium difficile infection. Am J Gastroenterol. 2012 Jul;107(7):1079-87. doi: 10.1038/ajg.2012.60. Epub 2012 Mar 27. PMID 22450732
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Carignan A, Poulin S, Martin P, Labbe AC, Valiquette L, Al-Bachari H, Montpetit LP, Pepin J. Efficacy of Secondary Prophylaxis With Vancomycin for Preventing Recurrent Clostridium difficile Infections. Am J Gastroenterol. 2016 Dec;111(12):1834-1840. doi: 10.1038/ajg.2016.417. Epub 2016 Sep 13. PMID 27619835
- [Background] Van Hise NW, Bryant AM, Hennessey EK, Crannage AJ, Khoury JA, Manian FA. Efficacy of Oral Vancomycin in Preventing Recurrent Clostridium difficile Infection in Patients Treated With Systemic Antimicrobial Agents. Clin Infect Dis. 2016 Sep 1;63(5):651-3. doi: 10.1093/cid/ciw401. Epub 2016 Jun 17. PMID 27318333